CLINICAL TRIAL: NCT04431362
Title: A Single Case Experimental Design Study Exploring the Effect of Music in an Inpatient Neuropsychological Rehabilitation Setting
Brief Title: Effects of Music Listening on Mood in an Inpatient Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 261210
Record Dates: First submitted 2019-04-26; First posted 2020-06-16 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants first complete a baseline phase before starting the intervention phase.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The measures will be completed by the clinical psychologist while the diary and checklist will be done by the patients with assistance from the research student or activity coordinators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Participants will not listen to music for 5 to 15 days based on the baseline duration they were assigned.
- Intervention (Experimental): Participants will listen to music for 3 weeks.
  Interventions: Behavioral: Self-selected music

INTERVENTIONS:
Behavioral: Self-selected music — Participants will be given iPods and headphones to listen to their music
  Arms: Intervention

SUMMARY:
The aim is to examine whether self-selected music can improve mood (as well as cognitive function) in stroke patients at an inpatient rehabilitation unit. Additionally, the feasibility of such an intervention will be assessed.

Hypotheses:

* The current intervention will be found to have a high feasibility.
* Stroke patients will exhibit improved mood during the music listening intervention phase compared to their baseline phase.
* Patients will show improvements in engagement in therapy if non-compliance was a previous issue (as demonstrated by therapist feedback regarding attendance of therapy sessions).
* Patients will experience improved cognitive (memory) function (i.e. immediate and delayed free recall) during the intervention phase compared to baseline.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of disability in the world. Research has shown that in the aftermath of a stroke, patients continue to experience various impairments even years after the stroke. For example, research has shown that stroke survivors continue to experience both cognitive impairments (e.g. executive dysfunction) and low mood (e.g. depression) even after more than 5 years since the stroke has passed. A further study was able to link low mood with reduced engagement in therapy, which has been found to lead patients to experience less benefits from the given therapy.

Due to the lack of supporting evidence for pharmacological and psychological treatments, music intervention was introduced with positive results being reported in regards to patients' mood and cognitive abilities. For example, one study found that stroke patients who listened to self-selected music were likely to experience a significant improvement in their mood and cognitive abilities when compared to another group who listened to audiobooks.

The current study aims to build on previous research by utilising a novel study design that has not been previously used to assess the feasibility and effectiveness of music intervention on the mood of patients located at an inpatient rehabilitation unit. The chosen design, single-case experimental design, allows researchers to take into account the individual differences of the patients, which cannot be considered when using an experimental design which needs a group of similar characteristics. In addition, by using a non-concurrent multiple baseline design, the researchers will be able to show that any changes occurring to the target behaviour (mood) will be due to the intervention itself rather than any other extraneous variables found in the environment, as three different time lengths will be used for the baseline phase (5, 10, and 15 days). The aim of the study is to provide data that support the feasibility and effectiveness of music intervention as an inexpensive and simple method for improving mood in stroke patients at an inpatient rehabilitation unit. It also aims to show similar effectiveness in increasing cognitive impairment and therapy engagement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Good grasp of the English Language
* Patients at the Frank Cooksey Rehabilitation Unit or transferring to the unit from an acute stroke ward
* Recent diagnosis of stroke using MRI or CT scans
* Low mood; will be confirmed by the clinical psychologist on the ward using mood screens as appropriate

Exclusion Criteria:- Severe or global aphasia, which interferes with their ability to understand instructions

* Have a diagnosis of dementia
* Patients who lack the capacity to consent

The study will also aim to exclude patients who have severe cognitive impairment, as assessed by the occupational therapists and clinical psychologist on the ward using screens or functional assessment as appropriate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the CORE-10 mood screen | up to 6 weeks
  questionnaire measure of distress, functioning and risk
Change in self-report diary | up to 6 weeks
  will assess feasibility by examining how frequently the patients are listening to music
Change in self-report by therapists | up to 6 weeks
  Will help to assess patients' engagement in therapy before during and after intervention
Change in the Montreal Cognitive Assessment | up to 6 weeks
  Will help to explore changes in cognition before and after the intervention. Minimum value=0, maximum value=30, better scores mean better outcome.
Change in The Brain Injury Rehabilitation Trust Memory and Information Processing Battery (examines memory and information processing. Only the story recall subcategory will be used) | up to 6 weeks
  Will help to explore changes in cognition (memory) before and after the intervention Minimum value=0, maximum value=60. Better scores mean better outcome
Change in the Mood Likert Scale | up to 6 weeks
  Ad hoc scale made for the study for participants to rate their mood. It is a Likert scale (0 is very relaxed, 10 is very stressed). Higher score thus mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Bellesi, DClinPsy, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamson J, Beswick A, Ebrahim S. Is stroke the most common cause of disability? J Stroke Cerebrovasc Dis. 2004 Jul-Aug;13(4):171-7. doi: 10.1016/j.jstrokecerebrovasdis.2004.06.003. PMID 17903971
- [Background] Dallery J, Cassidy RN, Raiff BR. Single-case experimental designs to evaluate novel technology-based health interventions. J Med Internet Res. 2013 Feb 8;15(2):e22. doi: 10.2196/jmir.2227. PMID 23399668
- [Background] Hammond MF, O'Keeffe ST, Barer DH. Development and validation of a brief observer-rated screening scale for depression in elderly medical patients. Age Ageing. 2000 Nov;29(6):511-5. doi: 10.1093/ageing/29.6.511. PMID 11191243
- [Background] Koorenhof L, Baxendale S, Smith N, Thompson P. Memory rehabilitation and brain training for surgical temporal lobe epilepsy patients: a preliminary report. Seizure. 2012 Apr;21(3):178-82. doi: 10.1016/j.seizure.2011.12.001. Epub 2011 Dec 23. PMID 22197200
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Ouellet MC, Morin CM. Efficacy of cognitive-behavioral therapy for insomnia associated with traumatic brain injury: a single-case experimental design. Arch Phys Med Rehabil. 2007 Dec;88(12):1581-92. doi: 10.1016/j.apmr.2007.09.006. PMID 18047872
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. Aphasiology. 2016 Jul 2;30(7):862-876. doi: 10.1080/02687038.2016.1178022. Epub 2016 Apr 29. PMID 27279674
- [Background] Tunnard C, Wilson BA. Comparison of neuropsychological rehabilitation techniques for unilateral neglect: an ABACADAEAF single-case experimental design. Neuropsychol Rehabil. 2014;24(3-4):382-99. doi: 10.1080/09602011.2013.872041. Epub 2014 Jan 13. PMID 24410191
- [Result] Ayerbe L, Ayis S, Wolfe CD, Rudd AG. Natural history, predictors and outcomes of depression after stroke: systematic review and meta-analysis. Br J Psychiatry. 2013 Jan;202(1):14-21. doi: 10.1192/bjp.bp.111.107664. PMID 23284148
- [Result] Baylan S, McGinlay M, MacDonald M, Easto J, Cullen B, Haig C, Mercer SW, Murray H, Quinn TJ, Stott D, Broomfield NM, Stiles C, Evans JJ. Participants' experiences of music, mindful music, and audiobook listening interventions for people recovering from stroke. Ann N Y Acad Sci. 2018 May 4. doi: 10.1111/nyas.13618. Online ahead of print. PMID 29727009
- [Result] Baylan S, Swann-Price R, Peryer G, Quinn T. The effects of music listening interventions on cognition and mood post-stroke: a systematic review. Expert Rev Neurother. 2016 Nov;16(11):1241-1249. doi: 10.1080/14737175.2016.1227241. Epub 2016 Aug 29. PMID 27548875
- [Result] Cumming TB, Churilov L, Linden T, Bernhardt J. Montreal Cognitive Assessment and Mini-Mental State Examination are both valid cognitive tools in stroke. Acta Neurol Scand. 2013 Aug;128(2):122-9. doi: 10.1111/ane.12084. Epub 2013 Feb 21. PMID 23425001
- [Result] Maclean N, Pound P, Wolfe C, Rudd A. Qualitative analysis of stroke patients' motivation for rehabilitation. BMJ. 2000 Oct 28;321(7268):1051-4. doi: 10.1136/bmj.321.7268.1051. PMID 11053175
- [Result] McKevitt C, Fudge N, Redfern J, Sheldenkar A, Crichton S, Rudd AR, Forster A, Young J, Nazareth I, Silver LE, Rothwell PM, Wolfe CD. Self-reported long-term needs after stroke. Stroke. 2011 May;42(5):1398-403. doi: 10.1161/STROKEAHA.110.598839. Epub 2011 Mar 24. PMID 21441153
- [Result] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Result] Skidmore ER, Whyte EM, Holm MB, Becker JT, Butters MA, Dew MA, Munin MC, Lenze EJ. Cognitive and affective predictors of rehabilitation participation after stroke. Arch Phys Med Rehabil. 2010 Feb;91(2):203-7. doi: 10.1016/j.apmr.2009.10.026. PMID 20159122
- See also: Neuro-rehabilitation beds open — http://www.kingshealthpartners.org/latest/629-neurorehabilitation-beds-open
- See also: Assessing capacity — http://www.nhs.uk/conditions/consent-to-treatment/capacity/
- See also: Frank Cooksey Rehabilitation Unit — http://www.kch.nhs.uk/service/a-z/frank-cooksey
- See also: Stroke — http://www.nhlbi.nih.gov/health-topics/stroke